CLINICAL TRIAL: NCT07346521
Title: Endoscopic Screening of Asymptomatic Patients for Helicobacter Pylori, Intestinal Metaplasia, and Barrett's Mucosa During Screening Colonoscopy - a Cross-sectional Study
Brief Title: Endoscopic Screening of Asymptomatic Patients for Helicobacter Pylori, Intestinal Metaplasia, and Barrett's Mucosa During Screening Colonoscopy
Acronym: G-SCOGE
Status: Recruiting | Type: Observational
Sponsor: Sigmund Freud PrivatUniversitat (Other)
Responsible Party: Sponsor
Other Study IDs: 17213538; 17213538 (Registry Identifier: Endoscopic screening of asymptomatic patients for H. pylori, IM, and Barrett's mucosa during Colonoscopy)
Record Dates: First submitted 2025-12-30; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: HELICOBACTER PYLORI INFECTIONS; Intestinal Metaplasia; Barett's Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asymptomatic patients undergoing Screening-Colonoscopy: A synchronous gastroscopy performed during colonoscopy at the patient's request to detect Helicobacter pylori infection.

SUMMARY:
The goal of this observational study is to learn how common Helicobacter pylori (H. pylori) infection is in adults without stomach or upper gastrointestinal symptoms who are having a preventive screening colonoscopy.

Endoscopic screening of the stomach is yet not acceptet as a standard screening procedure in Western countries. However, Helicobacter pylori infection is known to increase the risk of developing gastric cancer.

This study will look at the prevalence of Helicobacter pylori infection in asymptomatic patients who have an additional gastroscopy during the same session as their screening colonoscopy. It will also record other early tissue changes or risk factors for stomach cancer, such as intestinal metaplasia and Barrett's mucosa.

The main questions this study aims to answer are:

* How often is Helicobacter pylori found in adults without upper gastrointestinal symptoms by use of OGD?
* Are there any correlations between H. pylori infection and other risk factors, such as BMI, smoking, alcohol consumption, or a family history of colorectal and/or stomach cancer?

About 1000 participants are expected to take part. Adults undergoing a screening colonoscopy at a private endoscopy center will be offered the chance to have an additional gastroscopy if they meet the study's inclusion criteria (no previous Helicobacter pylori infection and no upper gastrointestinal symptoms).

Small tissue samples (biopsies) will be taken from the stomach and lower esophagus during the gastroscopy. Biopsies will be checked histologically for the presence of Helicobacter pylori and early tissue changes.

During the gastroscopy, no additional procedures or biopsies will be done beyond what is normally performed during a routine examination. Everything done during this procedure follows the standard steps of a regular gastroscopy.

All data will be coded to protect participant privacy. Researchers will use statistical methods to find out how common Helicobacter pylori infection is and whether it is related to other lifestyle or family risk factors or tissue changes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 30 years
* Scheduled screening colonoscopy (either initial screening or surveillance following previously detected polyps)
* Asymptomatic (no gastrointestinal symptoms)
* Willingness and consent to undergo simultaneous gastroscopy with biopsy sampling
* Written informed consent to participate in the study, including the use of histological findings and patient data for study analysis

Exclusion Criteria:

* Known Helicobacter pylori infection or previous treatment for H. pylori
* Current or recent proton pump inhibitor (PPI) therapy (< 4 weeks)
* Pre-existing gastrointestinal diseases (e.g., chronic gastritis, ulcer, gastric carcinoma)
* Immunosuppression or relevant underlying diseases
* Refusal to undergo additional gastroscopy or biopsy

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asymptomatic patients without upper gastrointestinal symptoms undergoing a Screening-Colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2026-12-16 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
The number of asymptomatic patients who are Helicobacter-positive. | From enrollment to the end of observation at 7 days
  All study participants undergo upper gastrointestinal endoscopy (gastroscopy). During the procedure, gastric biopsy specimens are obtained and subsequently processed for histopathological evaluation. The biopsies are analyzed to determine the presence of Helicobacter pylori infection. For statistical analysis, Helicobacter pylori status is coded as follows: absence of infection is recorded as 0, mild infection as 1, moderate infection as 2, and severe infection as 3.

SECONDARY OUTCOMES:
Asymptomatic patients who exhibit intestinal metaplasia and/or Barrett's mucosa. | From enrollment to the end of observation at 7 days
  During gastroscopy, biopsy specimens are obtained according to standard endoscopic protocols. Gastric biopsies are histopathologically processed and evaluated for the presence of intestinal metaplasia and Barrett's esophagus. Biopsies obtained from the stomach (Sydney Biopsie Protocol) the ora serrata are likewise histologically examined to identify the presence of Barrett's esophagus and/or intestinal metaplasia.The overall objective of this analysis is to assess the correlation, as well as the strength of the association, between the primary outcome, Helicobacter pylori infection, and the secondary outcomes, namely intestinal metaplasia and Barrett's mucosa.

OTHER OUTCOMES:
Association of BMI, smoking, alcohol consumption, and family history with gastric- and colorectal cancer in relation to Helicobacter pylori infection | From enrollment to the end of observation at 7 days
  The primary outcome of this study is the presence of Helicobacter pylori infection. Secondary outcome measures include potential risk factors such as body mass index (BMI), smoking, alcohol consumption, and family history of gastric and colorectal cancer, all evaluated in relation to Helicobacter pylori. BMI is calculated based on self-reported weight (in kilograms) and height (in meters) using the standard formula: BMI = weight / (height²). Alcohol consumption and smoking habits are recorded through participant self-report, as is family history, which is assessed by asking whether there is a documented occurrence of gastric or colorectal cancer in first-degree relatives. These measures allow the analysis of correlations between Helicobacter pylori infection and established risk factors

CONTACTS AND LOCATIONS:
Locations (1):
- Wiener Privatklinik (WPK), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Due to privacy regulations and restrictions of informed consent, de-identified individual participant data will not be made available.
  Additional Documents: Study protocol and statistical analysis plan may be provided upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: December 2025- December 2026 (12 months)